CLINICAL TRIAL: NCT03112005
Title: Assessment of EyeArt as an Automated Diabetic Retinopathy Screening Tool
Status: Completed | Type: Observational
Sponsor: Eyenuk, Inc. (Industry)
Collaborators: National Eye Institute (NEI) (NIH)
Responsible Party: Sponsor
Other Study IDs: EN-01; 9SB1EY027241 (NIH); 2R44EY026864 (NIH)
Record Dates: First submitted 2017-04-07; First posted 2017-04-13 (Actual); Last update posted 2018-07-30 (Actual); Status verified 2018-07

CONDITIONS: Diabetic Retinopathy; Diabetic Eye Problems; Diabetic Macular Edema
Keywords: Diabetic Eye Disease
MeSH Terms: conditions — Diabetic Retinopathy | interventions — Mydriatics

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

INTERVENTIONS:
Procedure: Color fundus photography — Subjects will undergo fundus photography before and after administration of mydriatic agent.
Drug: Mydriatic Agent — Subjects will be administered mydriatic medication to dilate their pupils.

SUMMARY:
More than 29 million people in the US are living with diabetes, many of whom will develop diabetic retinopathy (DR) or diabetic macular edema (DME) collectively known as diabetic eye disease (DED), the leading cause of vision loss and blindness in working-age adults. Annual eye screening is recommended for all diabetic patients since vision loss can be prevented with laser photocoagulation and anti-VEGF treatment if DR is diagnosed in its early stages. Currently, the number of clinical personnel trained for DR screening is orders of magnitude smaller than that needed to screen the large, growing diabetic population. Therefore, to meet this large unmet need for DR screening, a fully-automated computerized DR screening system is necessary.

EyeArt is an automated screening device designed automatically analyze color fundus photographs of diabetic patients to identify patients with referable or vision threatening DED. This study is designed to assess the safety and efficacy of EyeArt.

DETAILED DESCRIPTION:
This is a prospective, multi-center, observational study to assess the safety and efficacy of EyeArt in screening for DR.

This study will enroll up to 940 subjects who meet the eligibility criteria at eye care practices and primary/diabetes care practices. Subjects will undergo fundus photography per the EyeArt photography manual using commercially available, Food and Drug Administration (FDA) cleared, non-mydriatic fundus cameras.

Additionally, after dilation, the subject will undergo clinical reference standard photography by photographers certified to obtain photographs for clinical reference standard grading.

The EyeArt screening results on photographs obtained per the EyeArt photography manual will be compared with the clinical reference standard grading to evaluate the sensitivity and specificity of the EyeArt device.

The study will be conducted in accordance with applicable regulatory requirements and established rules for Good Clinical Practice (GCP). Study sites will be chosen to meet the study requirements.

Each study site will be visited periodically by the Study Monitor who will ascertain that all aspects of the Study Protocol are complied with and that the conduct of the study conforms to applicable regulatory requirements and established GCP rules.

At the time of each monitoring visit, the Study Monitor will review the completed case report forms (CRFs) to ascertain that all items have been completed and that the data provided are accurate and obtained in the manner specified in the protocol.

The Study Monitor will also check that the data in the CRF are consistent with the clinical records (Source Data Verification) and that study results are recorded completely and correctly. The Study Monitor will check on the reporting of adverse events (AEs).

All subject data will be captured utilizing a 21 CFR Part 11 compliant database. Electronic case report forms (eCRFs) will be source document verified by designated study monitors. Data entry of subject data will be performed by approved trained Site Personnel. Approved Site Personnel will have a user specific log-in name and password to access the electronic data capture (EDC) system in order to enter study data.

The EyeArt device will be finalized and frozen before the first subject is enrolled and a copy will be placed in a version-controlled system. Evidence that Eyenuk does not have direct access to the study data before data lock will include documentation, logs, and audit reports.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of diabetes mellitus;
* Understanding of study and provision of written informed consent; and
* 18 years of age or older.

Exclusion Criteria:

* Persistent visual impairment in one or both eyes;
* History of macular edema or retinal vascular (vein or artery) occlusion;
* History of ocular injections, laser treatment of the retina, or intraocular surgery other than cataract surgery without complications;
* Subject is contraindicated for fundus photography (for example, has light sensitivity);
* Subject has contraindications for mydriatic medications or is unwilling or unable to dilate;
* Subject is currently enrolled in an interventional study of an investigational device or drug; or
* Subject has a condition or is in a situation which in the opinion of the Investigator, might confound study results, may interfere significantly with the subject's participation in the study, or may result in ungradable clinical reference standard photographs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study subjects will be enrolled at eye care practices and primary/diabetes care practices
Sampling Method: Non-Probability Sample
Enrollment: 942 (Actual)
Dates: Start 2017-04-17 (Actual); Primary Completion 2018-05-31 (Actual); Study Completion 2018-05-31 (Actual)

PRIMARY OUTCOMES:
Number of subject eyes whose EyeArt results match the reading center grading for identifying referable diabetic eye disease (moderate NPDR or higher on the ICDR scale or surrogate markers for CSME). | 1 visit (1 day)
  The performance of EyeArt will be evaluated using sensitivity and specificity measures.
Number of subject eyes whose EyeArt results match the reading center grading for identifying vision threatening diabetic eye disease (severe NPDR or PDR or surrogate markers for CSME). | 1 visit (1 day)
  The performance of EyeArt will be evaluated using sensitivity and specificity measures.

CONTACTS AND LOCATIONS:
Locations (1):
- Los Angeles Biomedical Research Institute, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Undecided